CLINICAL TRIAL: NCT05747014
Title: Novapak Prospective Observational Clinical Trial
Acronym: Novapak
Status: Completed | Type: Observational
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT 22031
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Nasal Airway Obstruction
MeSH Terms: conditions — Nasal Obstruction | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Novapak Subjects: Subjects that are enrolled in the Novapak Study.
  Interventions: Device: Novapak Nasal Sinus Packing and Stent

INTERVENTIONS:
Device: Novapak Nasal Sinus Packing and Stent — Potential subjects will have the need to undergo nasal/sinus surgery using a space-occupying stent and will perform daily self-saline nasal irrigations.

SUMMARY:
The Novapak study is a prospective, observational, multi-site, non-controlled, non-randomized, case-series, with a 2 week and 1-month follow-up in adults undergoing nasal/sinus surgery with Novapak Nasal Sinus Packing and Stent device used as indicated post-operatively and is being conducted to obtain clinical data on the safety and effectiveness of the Novapak device under use as intended in the device indications.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of the Novapak Nasal Sinus Packing and Stent device used as indicated post-operatively in patients undergoing nasal/sinus surgery by:

* Collecting all AEs directly attributed to the device and/or those that cannot be determined; and calculating a point estimate and confidence interval
* Collecting all AEs and calculating an overall rate and safety profile for the device

The secondary objectives are to confirm device effectiveness through assessing adhesions, bleeding, healing and health during the procedure, 2 weeks and 1-month post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject undergoing nasal/sinus surgery with the intended need for nasal sinus packing (i.e., Novapak).
3. After being informed of the nature of the study; the subject understands, agrees to its provisions, is willing to participate and provide written consent.
4. Mentally stable and able to follow the instructions for self-assessment/questionnaire completion.

Exclusion Criteria:

1. Subject has a shellfish allergy.
2. Subject has known bleeding disorder or prescribed anticoagulants.
3. Subject has craniofacial abnormalities that may interfere with access to the sinuses.
4. Subject is immunocompromised (e.g., taking immunosuppressive medication).
5. Subject is participating in another investigational device, biologic, or drug study and has not completed the primary endpoint(s) or if there is a potential for clinical interference beyond the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the practices and clinics of the participating Study Investigators or from other non-investigator Otolaryngologist or Rhinologist physician referrals. Potential subjects will have the need to undergo nasal/sinus surgery using a space-occupying stent.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen R McKenzie, MS, Study Director — Medtronic
Locations (4):
- United States (3):
  - ENT Associates of South Florida, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
- St. Joseph's Health Care, London, Onterio, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | Novapak Subjects
Started (86 subjects consented to participate) | 86
Completed (77 subjects received Novapak implant) | 77
Not Completed | 9
Period: 14-Day Follow-up
Arm/Group | Novapak Subjects
Started | 77
Completed | 76
Not Completed | 1
Period: 30-Day Follow-up
Arm/Group | Novapak Subjects
Started | 76
Completed | 74
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Novapak Subjects
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.62 (17.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race was not collected for Canadian site. Only US sites were able to report race (n=57).
  Participants
    RACE: number analyzed (Participants) | 57
    RACE: WHITE | 40
    RACE: LATIN AMERICAN | 4
    RACE: NOT REPORTED | 2
    RACE: WHITE CARIBBEAN | 2
    RACE: AFRICAN AMERICAN | 1
    RACE: ARAB | 1
    RACE: ASIAN | 1
    RACE: ASIAN INDIAN | 1
    RACE: BAHAMIAN | 1
    RACE: BLACK OR AFRICAN AMERICAN | 1
    RACE: MEDITERRANEAN | 1
    RACE: MIDDLE EASTERN | 1
    RACE: OTHER | 1
Region of Enrollment [Number; unit: participants]
  Canada | 29
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessment - Adverse Events Related to Device
Description: Outcome Measure #1 for the Primary Outcome is the total number of Adverse Events that are directly attributed to the device and/or those that cannot be determined.
Time Frame: 30 days
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Groups:
- Total Number of Adverse Events Directly Attributed to the Device and/or Cannot be Determined: Total number of adverse events recorded that are attributed to the device or could not be determined.
  Novapak Nasal Sinus Packing and Stent: Potential subjects will have the need to undergo nasal/sinus surgery using a space-occupying stent and will perform daily self-saline nasal irrigations.
Arm/Group | Total Number of Adverse Events Directly Attributed to the Device and/or Cannot be Determined
Number analyzed (Participants) | 77
Number analyzed (Adverse Events) | 62
Adverse Events
  Device Relatedness - Causal Relationship | 0
  Device Relatedness - Probable | 1
  Device Relatedness - Possible | 2
  Device Relatedness - Not Related | 59

2. Primary Outcome: Safety Assessment - All Adverse Events
Description: Outcome Measure #2 for the Primary Outcome is the total number of Adverse Events.
Time Frame: 30 days
Measure: Number; unit: Adverse Events
Arm/Group | Novapak Subjects
Number analyzed (Participants) | 77
Adverse Events | 62

3. Secondary Outcome: Effectiveness Assessment - Total Number of Adhesions at Day 14 and Day 30 Post Treatment
Description: Outcome Measure #3 for the Secondary Outcome Measures is number of adhesions observed by endoscopic examination from procedure through 1-month post treatment.
Time Frame: 30 days
Population: This outcome was analyzed by sinus not by subject
Measure: Count of Units; unit: Sinuses
Units Other Than Participants: Sinuses
Groups:
- 14-Day Follow-up: Subjects that are enrolled in the Novapak Study and have completed their 14-day follow-up visit.
- 30-Day Follow-up: Subjects that are enrolled in the Novapak Study and have completed their 30-day follow-up visit.
Arm/Group | 14-Day Follow-up | 30-Day Follow-up
Number analyzed (Participants) | 76 | 74
Number analyzed (Sinuses) | 138 | 132
Sinuses | 6 | 5

4. Secondary Outcome: Effectiveness Assessment - Adhesion Grade at Day 14 and Day 30 Post Treatment
Description: Outcome Measure #4 for the Secondary Outcome Measures is the graded percentage of vertical height of the middle turbinate taken up by the adhesion using an ordinal scale (0-3), where '0' is No Adhesion Present, and '3' is >50% of middle turbinate height. This scoring is the Valentine method, and participants are graded based on their endoscopic examination.
Time Frame: 30 days
Population: For this outcome, analysis was done by sinus not by subject
Measure: Count of Units; unit: Sinuses
Units Other Than Participants: Sinuses
Arm/Group | 14-Day Follow-up | 30-Day Follow-up
Number analyzed (Participants) | 76 | 74
Number analyzed (Sinuses) | 138 | 132
Sinuses
  NO ADHESION PRESENT | 132 | 127
  < 25% OF MIDDLE TURBINATE HEIGHT | 5 | 4
  BETWEEN 25 AND 50% OF MIDDLE TURBINATE HEIGHT | 0 | 1
  >50% OF MIDDLE TURBINATE HEIGHT | 1 | 0

5. Secondary Outcome: Effectiveness Assessment - Bleeding Control
Description: Outcome Measure #5 for the Secondary Outcome Measures is to measure control of bleeding by comparing Boezaart Surgical Field Grading Scale scores post operatively, prior to Novapak insertion and post Novapak insertion. The Boezaart scale grades bleeding from Grade 0: No Bleeding through Grade 5: Severe Bleeding.
Time Frame: 1 day
Population: For this outcome, analysis was done by sinus, not by subject
Measure: Count of Units; unit: Sinuses
Units Other Than Participants: Sinuses
Groups:
- Prior to Novapak Insertion: Boezaart Surgical Field Grading prior to Novapak Insertion
- Post Novapak Insertion: Boezaart Surgical Field Grading after Novapak Insertion
Arm/Group | Prior to Novapak Insertion | Post Novapak Insertion
Number analyzed (Participants) | 77 | 77
Number analyzed (Sinuses) | 139 | 139
Sinuses
  GRADE 0: NO BLEEDING (CADAVERIC CONDITIONS) | 8 | 86
  GRADE 1: SLIGHT BLEEDING - NO SUCTIONING REQUIRED | 76 | 53
  GRADE 2: SLIGHT BLEEDING - OCCASIONAL SUCTIONING REQUIRED | 29 | 0
  GRADE 3: SLIGHT BLEEDING - FREQUENT SUCTIONING REQUIRED; BLEEDING THREATENS SURGICAL FIELD A FEW ... | 23 | 0
  GRADE 4: MODERATE BLEEDING - FREQUENT SUCTIONING REQUIRED AND BLEEDING THREATENS SURGICAL FIELD D... | 3 | 0
  GRADE 5: SEVERE BLEEDING - CONSTANT SUCTIONING REQUIRED; BLEEDING APPEARS FASTER THAN CAN BE REMO... | 0 | 0

6. Secondary Outcome: Effectiveness Assessment - Healing
Description: Outcome Measure #6 for the Secondary Outcome Measures is to measure healing by comparing Lund-Kennedy scores before surgery and at 2 weeks and 1-month post treatment. The Lund-Kennedy Scoring minimum is 0 and maximum is 10, with higher scores indicating worse observed disease. The Lund-Kennedy grading system is as follows:
  Nasal Polyps 0 = none; 1 = confined to middle meatus; 2 = beyond middle meatus Discharge 0 = none; 1 = clear and thin; 2 = thick and purulent Edema 0 = absent; 1 = mild; 2 = severe Scarring 0 = absent; 1 = mild; 2 = severe Crusting 0 = absent; 1 = mild; 2 = severe Numerical values for each term are summed for each sinus analyzed; and mean averages are reported.
Time Frame: 30 day
Population: For this outcome, analysis was done by sinus not by subject
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Sinuses
Groups:
- Pre-Surgery: Lund-Kennedy Score prior to surgery
- 14-Day Follow-up: Lund-Kennedy Score at 14-day follow-up
- 30-Day Follow-up: Lund-Kennedy Score at 30-day follow-up
Arm/Group | Pre-Surgery | 14-Day Follow-up | 30-Day Follow-up
Number analyzed (Participants) | 77 | 76 | 74
Number analyzed (Sinuses) | 139 | 138 | 132
score on a scale | 3.27 (1.95) | 1.99 (1.28) | 1.09 (1.26)

7. Secondary Outcome: Effectiveness Assessment - Health Assessment
Description: Outcome Measure #7 for the Secondary Outcome Measures is to measure health by comparing subject scores from the SNOT-22 questionnaire before surgery and at 2 weeks and 1-month post treatment. The Sino-Nasal Outcome Test (SNOT-22) is a validated questionnaire used to assess the severity of 22 symptoms related to the nasal sinuses using a 0-5-point scale (0 = No problem; 1 = Very mild problem; 2 = Mild or slight problem; 4 = Moderate problem; 5 = Problem as bad as it can be). Minimum score: 0; Maximum score: 110. The higher the score the worse the problems are.
Time Frame: 30 day
Population: The analysis population is number of subjects that completed the SNOT-22 questionnaire at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-Surgery: SNOT-22 Score prior to surgery
- 14-Day Follow-up: SNOT-22 Score at 14-day follow-up
- 30-Day Follow-up: SNOT-22 Score at 30-day follow-up
Arm/Group | Pre-Surgery | 14-Day Follow-up | 30-Day Follow-up
Number analyzed (Participants) | 79 | 75 | 72
score on a scale | 40.59 (18.05) | 25.03 (18.83) | 18.67 (16.80)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from procedure through 30-day follow-up.
Description: All adverse events that occurred from procedure through each subject's 30-day follow-up visit were collected.
Groups:
- Novapak Subjects: 86 total subjects were enrolled in the Novapak Study with 0 reported deaths. 77 subjects were implanted with the Novapak device and underwent Adverse Event Assessment(s).
  Novapak Nasal Sinus Packing and Stent: Potential subjects will have the need to undergo nasal/sinus surgery using a space-occupying stent and will perform daily self-saline nasal irrigations.
Arm/Group | Novapak Subjects
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 2/77
Other Adverse Events (participants affected / at risk) | 38/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novapak Subjects (N=77)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novapak Subjects (N=77)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Eye disorder (Eye disorders) | 1 (1)
Facial discomfort (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 (1)
Hyposmia (Nervous system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Scab (Skin and subcutaneous tissue disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Sinusitis bacterial (Infections and infestations) | 6 (6)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish as long as publications are provided to Medtronic for review at least 60 days prior to submission or presentation. Additionally, PIs will not independently publish, publicly disclose, present or discuss any Study results until a multi-center publication is released. If a multi-center publication is not released within one year after completion PIs will have the right to publish the results of and information pertaining to their activities on the Study.

DOCUMENTS (2):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT05747014/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT05747014/SAP_001.pdf